CLINICAL TRIAL: NCT06500884
Title: A Phase 2, Open-label, Randomized Study to Evaluate Prophylactic Interventions on Talquetamab-related Oral Toxicity
Brief Title: A Study to Evaluate Preventive Treatments for Talquetamab-related Oral Toxicity
Acronym: Talisman
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64407564MMY2006; 64407564MMY2006 (Other: Janssen Research & Development, LLC); 2023-506260-14-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Talquetamab (Active Comparator): Participants with relapsed or refractory multiple myeloma (RRMM) who are triple-class exposed (previously exposed to at least 1 proteasome inhibitor [PI], 1 immunomodulatory drug(s) [IMiD]), and an anti-CD38 monoclonal antibody [mAb]) will be treated with talquetamab subcutaneously until disease progression, death, unacceptable toxicity, withdrawal of consent, discontinuation of talquetamab, or end of study, whichever occurs first.
  Interventions: Drug: Talquetamab
- Cohort B: Prophylaxis A and Talquetamab (Experimental): Participants with RRMM who are triple-class exposed (previously exposed to at least 1 PI, 1 IMiD, and an anti-CD38 mAb) will receive prophylaxis A along with talquetamab therapy. Participants will start the assigned prophylaxis 7 days before starting talquetamab treatment. After step-up dosing of talquetamab therapy, participants will be treated with talquetamab with prophylaxes for up to 12 months during prophylaxis treatment phase (if there are clinical benefits prophylaxis treatment can continue beyond 12 months, at the treating physician's discretion, after consultation with sponsor). The Talquetamab treatment phase will continue from Cycle 1 Day 1 (C1D1) until disease progression, death, unacceptable toxicity, withdrawal of consent, discontinuation of talquetamab, or end of study, whichever occurs first.
  Interventions: Drug: Talquetamab; Drug: Prophylaxis A
- Cohort C: Prophylaxis B and Talquetamab (Experimental): Participants with RRMM who are triple-class exposed (previously exposed to at least 1 PI, 1 IMiD, and an anti-CD38 mAb) will receive prophylaxis B along with talquetamab therapy. Participants will start the assigned prophylaxis 7 days before starting talquetamab treatment. After step-up dosing of talquetamab therapy, participants will be treated with talquetamab with prophylaxes for up to 12 months during prophylaxis treatment phase (if there are clinical benefits prophylaxis treatment can continue beyond 12 months, at the treating physician's discretion, after consultation with sponsor). The Talquetamab treatment phase will continue from C1D1 until disease progression, death, unacceptable toxicity, withdrawal of consent, discontinuation of talquetamab, or end of study, whichever occurs first.
  Interventions: Drug: Talquetamab; Drug: Prophylaxis B
- Cohort D: Prophylaxis C and Talquetamab (Experimental): Participants with RRMM who are triple-class exposed (previously exposed to at least 1 PI, 1 IMiD, and an anti-CD38 mAb) will receive prophylaxis C along with talquetamab therapy. Participants will start the assigned prophylaxis 7 days before starting talquetamab treatment. After step-up dosing of talquetamab therapy, participants will be treated with talquetamab with prophylaxes for up to 12 months during prophylaxis treatment phase (if there are clinical benefits prophylaxis treatment can continue beyond 12 months, at the treating physician's discretion, after consultation with sponsor). The Talquetamab treatment phase will continue from C1D1 until disease progression, death, unacceptable toxicity, withdrawal of consent, discontinuation of talquetamab, or end of study, whichever occurs first.
  Interventions: Drug: Talquetamab; Drug: Prophylaxis C

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564
Drug: Prophylaxis A — Prophylaxis A will be administered orally.
  Arms: Cohort B: Prophylaxis A and Talquetamab
Drug: Prophylaxis B — Prophylaxis B will be administered orally.
  Arms: Cohort C: Prophylaxis B and Talquetamab
Drug: Prophylaxis C — Prophylaxis C will be administered orally.
  Arms: Cohort D: Prophylaxis C and Talquetamab

SUMMARY:
The purpose of this study is to identify preventive treatments that can minimize the occurrence, severity, and duration of talquetamab-related taste changes (dysgeusia), during the prophylaxis (preventive) treatment phase, and to better characterize the signs or symptoms of talquetamab-related taste changes.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma (MM) according to IMWG diagnostic criteria
* Were triple-class exposed (received prior treatment with a PI, an IMiD, and anti CD38 mAb)
* Documented evidence of progressive disease based on investigator's determination of response by IMWG criteria on or after their last regimen
* Have an Eastern Cooperative Oncology Group-performance status (ECOG-PS) of 0 or 1 at screening. Participants with ECOG-PS 2 or 3 are eligible for the study if the ECOG-PS score is related to stable physical limitations (e.g., wheelchair-bound due to prior spinal cord injury) and not related to multiple myeloma or associated therapy
* Be willing and able to adhere to the lifestyle restrictions specified in the protocol

Exclusion Criteria:

* Contraindications or life-threatening known allergies, hypersensitivity, or intolerance to any study drug or its excipients
* Stroke, transient ischemic attack, or seizure within 6 months prior to screening
* Any of the following within 6 months prior to the first dose of study treatment: severe or unstable angina, myocardial infarction; major thromboembolytic event (e.g., pulmonary embolism, cerebrovascular accident), clinically significant ventricular arrythmia or heart failure New York Heart Association functional classification Class III or IV. Uncomplicated deep vein thrombosis is not considered exclusionary
* Major surgery or had significant traumatic injury within 2 weeks prior to the start of administration of talquetamab, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment
* A WETT score suggesting severe dysgeusia at screening. Also unresolved/severe dysgeusia referred by the participant or a finding in the physical examination/oral cavity inspection. Some examples include leukoplakia, prior mouth cancers, extensive dental caries, severe periodontitis, active oral infections, candidiasis, parotic gland removal, or radiotherapy with resultant xerostomia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Occurrence of Dysgeusia as Assessed by the Total Waterless Empirical Taste Test (WETT) Testing Score During the Prophylaxis Treatment Phase | Up to 12 months
  Dysgeusia is defined as total WETT score of 25th percentile or below according to the Normative WETT-SA53 percentile table. Taste assessment will be performed using taste strips (WETT). Four concentrations (4=lowest concentration, 1=highest concentration) will be used for each taste quality: sweet, sour, salty, bitter, and umami. Each test kit contains 53 taste strips distributed in 4 packs; and each taste strip is numbered (1 through 53). Participants will use each strip sequentially and record the flavor on a score card provided. The test will result in a maximum (that is, best) total score of 53. The score will be graded by a qualified site staff into a normative percentile score using a provided chart.
Percentage of Participants With Occurrence of Severe Dysgeusia During the Prophylaxis Treatment Phase | Up to 12 months
  Severe Dysgeusia is defined as a total WETT score of 10th percentile or below according to the normative WETT-SA53 percentile table. Taste assessment will be performed using taste strips (WETT). Four concentrations (4=lowest concentration, 1=highest concentration) will be used for each taste quality: sweet, sour, salty, bitter, and umami. Each test kit contains 53 taste strips distributed in 4 packs; and each taste strip is numbered (1 through 53). Participants will use each strip sequentially and record the flavor on a score card provided. The test will result in a maximum (that is, best) total score of 53. The score will be graded by a qualified site staff into a normative percentile score using a provided chart.
Time to the First Onset of Severe Dysgeusia During the Prophylaxis Treatment Phase | Up to 12 months
  Time to the first onset of severe dysgeusia is defined as time from the first dose date of talquetamab to the first onset date of severe dysgeusia according to the total WETT score. Taste assessment will be performed using taste strips (WETT). Four concentrations (4=lowest concentration, 1=highest concentration) will be used for each taste quality: sweet, sour, salty, bitter, and umami. Each test kit contains 53 taste strips distributed in 4 packs; and each taste strip is numbered (1 through 53). Participants will use each strip sequentially and record the flavor on a score card provided. The test will result in a maximum (that is, best) total score of 53. The score will be graded by a qualified site staff into a normative percentile score using a provided chart.
Percentage of Participants Who Report Resolution/Improvement of Dysgeusia During the Prophylaxis Treatment Phase | At Month 3
  Resolution/improvement is defined as 2 potential scenarios: 1) A dysgeusia downgraded to dysgeusia-free, that is (i.e.,) total WETT score of 25th percentile or below at visits prior to the end of month 3 becomes total WETT score above 25th percentile at the end of month 3. 2) Severe dysgeusia downgraded to non-severe dysgeusia, i.e., total WETT score of 10th percentile or below prior to the end of month 3 becomes total WETT score above 10th percentile at the end of month 3. Taste assessment will be performed using taste strips (WETT). Four concentrations will be used for each taste quality: sweet, sour, salty, bitter, & umami. Each test kit contains 53 taste strips; numbered (1 through 53). Participants will use each strip sequentially and record flavor on score card provided. Test will result in maximum (i.e., best) total score of 53. Score will be graded by qualified staff into normative percentile score using provided chart.
Percentage of Participants Who Report Resolution/Improvement of Dysgeusia During the Prophylaxis Treatment Phase | At Month 6
  Resolution/improvement is defined as 2 potential scenarios: 1) A dysgeusia downgraded to dysgeusia-free, that is (i.e.,) total WETT score of 25th percentile or below at visits prior to the end of month 6 becomes total WETT score above 25th percentile at the end of month 6. 2) Severe dysgeusia downgraded to non-severe dysgeusia, i.e., total WETT score of 10th percentile or below prior to the end of month 6 becomes total WETT score above 10th percentile at the end of month 6. Taste assessment will be performed using taste strips (WETT). Four concentrations will be used for each taste quality: sweet, sour, salty, bitter, & umami. Each test kit contains 53 taste strips; numbered (1 through 53). Participants will use each strip sequentially and record flavor on score card provided. Test will result in maximum (i.e., best) total score of 53. Score will be graded by qualified staff into normative percentile score using provided chart.

SECONDARY OUTCOMES:
Change From Baseline in WETT Testing Score Over Time | Baseline up to 30 months
  Taste assessment will be performed using taste strips (WETT). Four concentrations (4=lowest concentration, 1=highest concentration) will be used for each taste quality: sweet, sour, salty, bitter, and umami. Each test kit contains 53 taste strips distributed in 4 packs; and each taste strip is numbered (1 through 53). Participants will use each strip sequentially and record the flavor on a score card provided. The test will result in a maximum (that is, best) total score of 53.
Percentage of Time with Dysgeusia During the Prophylaxis Treatment Phase | Up to 12 months
  Time with dysgeusia is defined as the accumulative days a participant had dysgeusia according to the total WETT score divided by the total days of talquetamab exposure. Taste assessment will be performed using taste strips (WETT). Four concentrations (4=lowest concentration, 1=highest concentration) will be used for each taste quality: sweet, sour, salty, bitter, and umami. Each test kit contains 53 taste strips distributed in 4 packs; and each taste strip is numbered (1 through 53). Participants will use each strip sequentially and record the flavor on a score card provided. The test will result in a maximum (that is, best) total score of 53. The score will be graded by a qualified site staff into a normative percentile score using a provided chart.
Number of Participants with Treatment-emergent Oral Toxicities (Dysgeusia, Oral Mucositis, Dysphagia, and Xerostomia) During the Prophylaxis Treatment Phase | Up to 12 months
  Oral toxicity including dysgeusia, oral mucositis, dysphagia, and xerostomia will be graded (including Grade 0 for dysgeusia) based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 5.0. Severity has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; and Grade 5: Death.
Number of Participants with Treatment-emergent Oral Toxicities (Dysgeusia, Oral Mucositis, Dysphagia, and Xerostomia) Over Time | Up to 30 months
  Oral toxicity including dysgeusia, oral mucositis, dysphagia, and xerostomia will be graded (including Grade 0 for dysgeusia) based on NCI-CTCAE, Version 5.0. Severity has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; and Grade 5: Death.
Time to the First Onset of Treatment-emergent Oral Toxicities (Dysgeusia, Oral Mucositis, Dysphagia, and Xerostomia) | Up to 30 months
  Time to the first onset of treatment-emergent dysgeusia, oral mucositis, dysphagia, or xerostomia, will be summarized.
Duration of Treatment-emergent Oral Toxicities (Dysgeusia, Oral Mucositis, Dysphagia, and Xerostomia) | Up to 30 months
  Duration of treatment-emergent oral toxicities including dysgeusia, oral mucositis, dysphagia, and xerostomia will be reported in this outcome measure.
Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 items (EORTC-QLQ-C30) Domains Scores Over Time | From Baseline up to 30 months
  The EORTC-QLQ-C30 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days, and responses are reported using verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high health related quality of life (HRQoL), but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Oral Health (EORTC-QLQ-OH15) Domains Scores Over Time | From Baseline up to 30 months
  The EORTC module QLQ-OH15 is a 15-item, well-accepted, and validated assessment tool focusing on oral problems and quality of life. The recall period for symptoms is 7 days and response options include 'not at all', "a little', 'quite a bit', and 'very much'. All of the items' measures range in score from 0 to 100. A high score for the symptom items represents a high level of symptomatology or problems.
Percentage of Participants Reporting Oral Symptoms Using the Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 12 months
  PRO-CTCAE is a patient-reported item custom survey used to evaluate symptomatic treatment-emergent adverse events in participants on cancer clinical trials. The PRO-CTCAE custom survey consists of 18 items. Responses are provided on a 5-point Likert scale that ranges from 0 to 4. The recall period for symptoms is 7 days. Higher scores indicating greater severity/impact.
Percentage of Participants Reporting Oral Symptoms Using the Short Xerostomia Inventory (SXI) Score | Up to 30 months
  SXI is a validated questionnaire that explores how the participant experiences dry mouth (xerostomia) with 5 questions extracted from the original XI. Respondents are asked to choose 1 of 5 responses ("1-Never; 2-Hardly ever; 3-Occasionally; 4-Fairly often; and 5-Very often") to specific statements referring to the preceding 4 weeks. Each individual's responses are scored and summed to give a single XI score. Higher scores represent more severe symptoms.
Percentage of Participants Reporting Oral Symptoms Using the Epstein Taste Survey (ETS) | Up to 30 months
  The Epstein Taste Survey (ETS) consists of 17 items PRO instrument, specific to taste and smell changes. The ETS was developed for use in participants with head and neck cancer. This instrument will be used to measure treatment-related symptoms associated with talquetamab.
Percentage of Participants Reporting Oral Symptoms Using the Scale of Subjective Total Taste Acuity (STTA) | Up to 12 months
  The STTA is a tool to assess the overall acuity of taste based on a 4-point scale, where 0 reflects no change and 4 represents almost complete loss of taste function. Higher score indicating severity.
Change from Baseline in Body Weight Over Time | From Baseline up to 30 months
  Change from baseline in body weight will be reported.
Change from Baseline in Body Mass Index (BMI) Over Time | From Baseline up to 30 months
  Change from baseline in BMI will be reported.
Percentage of Participants With Dose Reductions, Interruptions, and Discontinuations | Up to 12 months
  Percentage of participants with dose reductions, dose interruptions, and dose discontinuations will be reported.
Change from Baseline in Smell Identification Test Score | Baseline (Day 1 Cycle 1), Day 1 Cycle 2 (each cycle duration=28-days)
  Smell identification testing will be performed using 4 booklets each containing 10 labels that will release a distinctive scent when scraped with a pencil. Participants will choose the appropriate scent from the associated options. The minimum possible score is a 0 and the maximum is a 40. A higher score indicates better smell/outcome.
Change from Baseline in Smell Detection Threshold Test Score | Baseline (Day 1 Cycle 1), Day 1 Cycle 2 (each cycle duration=28-days)
  Smell threshold detection testing will be performed using vials of rose oil (phenyl ethanol) in vol/vol concentrations ranging from 10^-2 (strongest) through 10^-9 (weakest). Participants will be exposed, one at a time, to pairs of vials and asked to distinguish which is stronger.
Percentage of Participants With Overall Response Rate | Up to 30 months
  Overall response rate is defined as the participants with a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.
Percentage of Participants With Complete Response (CR) or Better Response | Up to 30 months
  CR or better response is defined as the participants who achieve a CR or better response according to the IMWG criteria.
Percentage of Participants With Very Good Partial Response (VGPR) or Better Response | Up to 30 months
  VGPR or better response is defined as the percentage of participants who achieve a VGPR or better response according to the IMWG criteria.
Duration of Response (DOR) | Up to 30 months
  Duration of response is defined as time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria, or death due to disease progression, whichever occurs first.
Time to Response (TTR) | Up to 30 months
  Time to response is defined as the time between date of first dose of talquetamab and the first efficacy evaluation at which the participant has met all criteria for PR or better.
Progression-free Survival (PFS) | Up to 30 months
  PFS is defined as the time from the date of first dose of talquetamab to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Number of Participants with Treatment-emergent Adverse Event (TEAEs) | Up to 30 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study treatment through the day of last dose plus 30 days, or if beyond 30 days from last dose but is study treatment-related, is considered to be treatment-emergent.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (38):
- United States (9):
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Brazil (6):
  - Hospitais Integrados da Gavea SA DF Star, Brasília
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Hospital Erasto Gaertner- Liga Paranaense de Combate ao Cancer, Curitiba
  - Instituto D Or de Pesquisa e Ensino, Salvador
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
- Netherlands (3):
  - VUMC Amsterdam, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Erasmus MC, Rotterdam
- Hospital Espanol Auxilio Mutuo Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Virgen de La Arrixaca, El Palmar
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - Colchester Hospital University NHS, Colchester
  - Eastbourne District General Hospital, Eastbourne
  - The Clatterbridge Cancer Centre, Liverpool
  - University College London Hospitals, London
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Newcastle Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency